CLINICAL TRIAL: NCT02824705
Title: Effects of Cardiac ICU Practice Variation on Intestinal Epithelial Barrier Function and Microbiome Diversity
Brief Title: Kids Intestinal Dysfunction in Congenital Heart Disease: the Kind Heart Study
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Katri Typpo, Principal Investigator, University of Arizona
Other Study IDs: NIDDK
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Congenital Disease
Keywords: Heart; multiple organ dysfunction syndrome; pediatric critical care; congenital heart disease
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Multiple Organ Failure; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples, blood samples with permission of family
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Congenital Heart Disease Surgery — Stool and blood sample collected prior to surgical intervention for congenital heart disease; stool and blood samples then collected in days following cardiac intervention.

SUMMARY:
Approximately 40,000 infants are born each year in the United States with congenital heart defects (CHD), and heart defects are the leading cause of birth defect-related deaths in the United States. While advances in surgical treatment, cardiac bypass, and post-operative management have improved mortality for children born with heart defects, these children continue to have significant morbidity related to post-operative malnutrition, multiple organ dysfunction (MODS), and sepsis. Proposed mechanisms for post-operative sepsis and MODS is via loss of intestinal epithelial barrier function (EBF) or intestinal micro biome diversity.

The purpose of this multi-center observational cohort study is to understand the extent to which practice variation for routine post-operative care might worsen intestinal barrier dysfunction and reduce diversity of the intestinal microbiome for infants undergoing surgical correction of left sided cardiac obstructive defects. We will enroll 80 children with left sided obstructive congenital cardiac lesions across several US congenital cardiac centers to obtain clinical data and biological specimens. We will leverage existing differences in nutritional and antibiotic strategies at these centers to better understand how intestinal barrier function and the intestinal microbiome may contribute to post-operative multiple organ dysfunction syndrome.

ELIGIBILITY:
Inclusion Criteria:

* pre-operative diagnosis of left sided obstructive congenital cardiac defect

Exclusion Criteria:

* Corrected gestational age < 37 weeks at time of surgery
* Short bowel syndrome
* Intestinal graft vs. host disease
* Inflammatory Bowel Disease (Ulcerative Colitis, or Crohn's disease)
* Candidate for intestinal transplant
* History of necrotizing enterocolitis (NEC)
* Previous Randomization into this study

Ages: 3 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of infants and young children who are diagnosed with left sided obstructive congenital heart disease and are scheduled for corrective surgery. Investigators will enroll a total of 80 patients in this multi-center trial. Investigators anticipate that local enrollment will be about 1-2 patients per month, or 12-24 per year when the cardiac program is active.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2016-04; Primary Completion 2021-01-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline intestinal epithelial barrier biomarker profile | 04/2016-01/31/2020
Microbiome diversity | 04/2016-01/31/2020

SECONDARY OUTCOMES:
Multiple Organ Dysfunction Syndrome | 04/2016-01/31/2020

CONTACTS AND LOCATIONS:
Overall Officials: Katri Typpo, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No